CLINICAL TRIAL: NCT02144987
Title: New Therapeutic Approaches to Treat Asherman's Syndrome and Endometrial Atrophy Based in BM Stem Cells Autologous Transplantation
Brief Title: Bone Marrow Stem Cell Treatment for Asherman's Syndrome and Endometrial Atrophy
Acronym: BMSCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1101-C-092-JS
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Asherman's Syndrome; Endometrium; Atrophy, Cervix
MeSH Terms: conditions — Gynatresia; Atrophy | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Bone Marrow CD133+ Stem Cell Transplantation — 1. Bone Marrow Stem Cell (BMSC) mobilization peripheral blood induced by granulocyte-CSF (G-CSF) 5 mcg/kg sc every 12 hours for 4 days.
  2. BMSC recollection with apheresis procedure and positive selection of the CD133+ cells.
     The selection procedure will be performed for a maximum of 3 hours or until at least 50 million cells are collected.
  3. CD133+ cells transplantation into the uterine spiral arterioles by intra-arterial catheterization
  4. Subsequently Hormonal Replacement Therapy (HRT) will be given to the patients
  5. Hysteroscopy will be performed 2-3 months after stem cell transplantation
  6. Embryo transfer will be performed 3-6 months after stem cell transplantation with HRT endometrial preparation
  Other Names: Neupogen

SUMMARY:
The purpose of this study is to determine whether Bone Marrow Stem Cell transplantation may improve Assisted Reproduction Techniques (ART) outcomes in refractive Asherman's Syndrome or Atrophic Endometrium.

DETAILED DESCRIPTION:
This novel technique refers to the use of CD133+ autologous bone marrow stem-cells to regenerate the endometrium in patients with Asherman's Syndrome, Endometrial Atrophy or any condition that produce a destruction of the endometrium or its de novo creation in a bioengineered uterus.

It requires a previous mobilization in the peripheral blood of CD133+ autologous bone marrow stem cells, subsequent apheresis and transplant of the same cells in the spiral arterioles of the uterus with the aim to regenerate de novo the endometrium. This technique represents a new therapeutical approach for the treatment of endometrial regeneration problems such Asherman Syndrome and the endometrial atrophy since currently no specific treatment for these endometrial pathologies exist.

A prospective experimental non controlled study has been designed in order to assess the effectiveness of these technique as a new tool for treat Asherman's Syndrome and Endometrial Atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of Asherman Syndrome and absence of pregnancy after treatment
* Endometrial atrophy (<6mm) with Implantation Failure
* Age 20-45 years-old
* Normal liver, heart and kidney function
* Presence of menstrual bleeding with Natural Cycle or HRT
* Absence of psychiatric pathology and ability to accomplish the treatment
* β-hCG negative
* Absence of SDT

Exclusion Criteria:

* Absence of peripheral vein access
* Lack of accomplish inclusion criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Live-birth rate | 15 months
  Live birth rate is the percentage of all cycles that lead to live birth, and is the pregnancy rate adjusted for miscarriages and stillbirths.
Ongoing pregnancy rate | 9 months
  Ongoing pregnancy rate is the percentage of all cycles that lead to presence of heartbeat in Ultrasound scan at the end of the first trimester
Implantation Rate | 6 months
  Implantation rate is the percentage of embryos which successfully undergo implantation compared to the number of embryos transferred in a given period.

SECONDARY OUTCOMES:
Endometrial thickness prior to the treatment | 0
  Endometrial thickness measured with Ultrasound in a previous treatment with Hormonal Replacement Therapy
Endometrial Thickness after treatment | 3-6 months
  Endometrial thickness measured with Ultrasound with Hormonal Replacement Therapy 3-6 months after Bone Marrow Stem Cell Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Santamaria, MD, PhD, Principal Investigator — Instituto Valenciano Infertilidad; Carlos Simon, MD, PhD, Principal Investigator — Instituto Valenciano Infertilidad
Locations (2):
- Spain (2):
  - Hospital Clinico y Universitario de Valencia, Valencia, Valencia
  - Instituto Valenciano Infertilidad, Valencia, Valencia

REFERENCES:
- [Background] Chan RW, Schwab KE, Gargett CE. Clonogenicity of human endometrial epithelial and stromal cells. Biol Reprod. 2004 Jun;70(6):1738-50. doi: 10.1095/biolreprod.103.024109. Epub 2004 Feb 6. PMID 14766732
- [Background] Cervello I, Gil-Sanchis C, Mas A, Faus A, Sanz J, Moscardo F, Higueras G, Sanz MA, Pellicer A, Simon C. Bone marrow-derived cells from male donors do not contribute to the endometrial side population of the recipient. PLoS One. 2012;7(1):e30260. doi: 10.1371/journal.pone.0030260. Epub 2012 Jan 19. PMID 22276168
- [Background] Ikoma T, Kyo S, Maida Y, Ozaki S, Takakura M, Nakao S, Inoue M. Bone marrow-derived cells from male donors can compose endometrial glands in female transplant recipients. Am J Obstet Gynecol. 2009 Dec;201(6):608.e1-8. doi: 10.1016/j.ajog.2009.07.026. Epub 2009 Oct 3. PMID 19800602
- [Background] Taylor HS. Endometrial cells derived from donor stem cells in bone marrow transplant recipients. JAMA. 2004 Jul 7;292(1):81-5. doi: 10.1001/jama.292.1.81. PMID 15238594
- [Background] Cervello I, Mas A, Gil-Sanchis C, Peris L, Faus A, Saunders PT, Critchley HO, Simon C. Reconstruction of endometrium from human endometrial side population cell lines. PLoS One. 2011;6(6):e21221. doi: 10.1371/journal.pone.0021221. Epub 2011 Jun 21. PMID 21712999
- [Background] Nagori CB, Panchal SY, Patel H. Endometrial regeneration using autologous adult stem cells followed by conception by in vitro fertilization in a patient of severe Asherman's syndrome. J Hum Reprod Sci. 2011 Jan;4(1):43-8. doi: 10.4103/0974-1208.82360. PMID 21772740
- [Background] March CM. Management of Asherman's syndrome. Reprod Biomed Online. 2011 Jul;23(1):63-76. doi: 10.1016/j.rbmo.2010.11.018. Epub 2010 Dec 4. PMID 21549641
- [Background] Zhang X, Chen CH, Confino E, Barnes R, Milad M, Kazer RR. Increased endometrial thickness is associated with improved treatment outcome for selected patients undergoing in vitro fertilization-embryo transfer. Fertil Steril. 2005 Feb;83(2):336-40. doi: 10.1016/j.fertnstert.2004.09.020. PMID 15705371
- [Background] Sanz-Ruiz R, Gutierrez Ibanes E, Arranz AV, Fernandez Santos ME, Fernandez PL, Fernandez-Aviles F. Phases I-III Clinical Trials Using Adult Stem Cells. Stem Cells Int. 2010 Nov 4;2010:579142. doi: 10.4061/2010/579142. PMID 21076533
- [Background] Makela J, Anttila V, Ylitalo K, Takalo R, Lehtonen S, Makikallio T, Niemela E, Dahlbacka S, Tikkanen J, Kiviluoma K, Juvonen T, Lehenkari P. Acute homing of bone marrow-derived mononuclear cells in intramyocardial vs. intracoronary transplantation. Scand Cardiovasc J. 2009 Dec;43(6):366-73. doi: 10.1080/14017430903045350. PMID 19544220
- [Derived] Santamaria X, Cabanillas S, Cervello I, Arbona C, Raga F, Ferro J, Palmero J, Remohi J, Pellicer A, Simon C. Autologous cell therapy with CD133+ bone marrow-derived stem cells for refractory Asherman's syndrome and endometrial atrophy: a pilot cohort study. Hum Reprod. 2016 May;31(5):1087-96. doi: 10.1093/humrep/dew042. Epub 2016 Mar 22. PMID 27005892
- [Derived] Cervello I, Gil-Sanchis C, Santamaria X, Cabanillas S, Diaz A, Faus A, Pellicer A, Simon C. Human CD133(+) bone marrow-derived stem cells promote endometrial proliferation in a murine model of Asherman syndrome. Fertil Steril. 2015 Dec;104(6):1552-60.e1-3. doi: 10.1016/j.fertnstert.2015.08.032. Epub 2015 Sep 15. PMID 26384164